CLINICAL TRIAL: NCT00123292
Title: An Open-label, Ascending-dose, Clinical Trial of Intra-arterial Microplasmin Administration in Patients With Acute Peripheral Arterial Occlusion
Brief Title: Intra-arterial Microplasmin Administration in Patients With Acute Peripheral Arterial Occlusion
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision not to pursue development of uPLi for vascular conditions
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG-M-002
Record Dates: First submitted 2005-07-21; First posted 2005-07-22 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Arterial Occlusive Diseases
Keywords: arterial occlusion; thromboembolism; Acute Peripheral Arterial Occlusion
MeSH Terms: conditions — Arterial Occlusive Diseases; Thromboembolism | interventions — microplasmin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: Microplasmin
- 2 (Experimental)
  Interventions: Drug: Microplasmin
- 3 (Experimental)
  Interventions: Drug: Microplasmin
- 4a (Experimental)
  Interventions: Drug: Microplasmin
- 4b (Experimental)
  Interventions: Drug: Microplasmin

INTERVENTIONS:
Drug: Microplasmin — An infusion of 0.45, 0.60 and 0.90 mg/kg/hr will be administered for up to 4 hours. Study drug will be administered intra-arterially (into the thrombotic occlusion).
  Arms: 1; 2; 3
Drug: Microplasmin — An infusion of 0.45 mg/kg/hr in conjunction with distal protection device will be administered for up to 4 hours. Study drug will be administered intra-arterially (into the thrombotic occlusion).
  Arms: 4a
Drug: Microplasmin — An infusion of 20 or 40 mg (20 mg for the 15 cm treatment length device; 40 mg for the 30 cm treatment length device) over 10 minutes via the Trellis-8 Peripheral Infusion System catheter, in accordance with the Trellis-8 Instructions for Use. For occlusive lesions that are longer than the treatment length of the Trellis-8 device, a repeat infusion of the same dose and duration may be administered.
  Arms: 4b

SUMMARY:
The purpose of the trial is to evaluate the safety and efficacy of microplasmin administration in patients with acute peripheral arterial occlusion.

DETAILED DESCRIPTION:
This clinical trial is designed as an open-label, dose-escalating, single-centre trial of weight-adjusted dose regimens of microplasmin administered intra-arterially as an infusion to patients with acute peripheral arterial occlusion. Patients who meet all inclusion criteria and none of the exclusion criteria will be administered study drug for up to 4 hours. Different dose regimens will be evaluated in an ascending-dose fashion; an infusion will be administered for up to 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting within 14 days of onset of acute thrombotic or embolic arterial occlusion of a lower extremity (native vessel or bypass graft).
* Complete occlusion of infrarenal vessel or bypass graft, as determined by angiography.
* Lower extremity ischemia graded as SVS/ISCS (Society of Vascular Surgery/ International Society for Cardiovascular Surgery) class I or II (a or b).
* Negative urine pregnancy test (pregnancy test only required for females of child-bearing potential not using an accepted method of contraception).

Exclusion Criteria:

* Profound ischemia with permanent motor paresis or sensory loss (or ischemic process deemed irreversible, i.e. class III).
* Occlusion not penetrable by the infusion guide wire.
* Known or suspected allergy to contrast agents or heparin sodium.
* Active bleeding or known hemorrhagic diathesis.
* Stroke in the previous 6 months or transient ischemic attack in the previous 2 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-03; Primary Completion 2007-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Complete clot-lysis (defined as >95% estimated clot volume reduction compared to baseline angiogram) | at 4 hours or less (if study drug administration is terminated prior to 4 hours).

SECONDARY OUTCOMES:
Proportion of subjects with clot-lysis (complete or partial, defined as any clot volume reduction on angiography) | At 4 hours or less (if study drug administration is terminated prior to 4 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Peter Verhamme, MD, PhD, Principal Investigator — KU Leuven
Locations (1):
- University Hospital Gasthuisberg, Leuven, Belgium